CLINICAL TRIAL: NCT03721276
Title: Project EQuIP: Empowering Queer Identities in Psychotherapy
Acronym: EQuIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000020997; R01MH109413 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Sexual Minority Stress
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Masking Description: Patients will either be immediately enrolled or wait listed for the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy (Experimental): Individuals assigned to therapy will receive 10 weekly individually-delivered sessions, directly after baseline assessment, that address minority stress mechanisms underlying SMW's depression, anxiety, and alcohol abuse.
  Interventions: Behavioral: EQuIP (Empowering Queer Identities in Psychotherapy)
- Waitlist (Other): Individuals assigned to waitlist will be put on a waitlist for 3 months after baseline assessment, after which they will also receive the same treatment as the therapy group.
  Interventions: Behavioral: EQuIP (Empowering Queer Identities in Psychotherapy)

INTERVENTIONS:
Behavioral: EQuIP (Empowering Queer Identities in Psychotherapy) — Individuals assigned to therapy will receive 10 weekly individually-delivered sessions, directly after baseline assessment, that address minority stress mechanisms underlying SMW's depression, anxiety, and alcohol abuse.
  Other Names: ESTEEM (Effective Skills to Empower Effective Men) for Women

SUMMARY:
The aim of this study is to develop an evidence-based psychosocial intervention for sexual minority women. This intervention will specifically target the adverse mental and behavioral health outcomes disproportionately experienced by sexual minority women, including depression, suicidality, and alcohol abuse, which are known to be driven by stigma-related stressors associated with their sexual orientation (i.e., minority stress processes).

DETAILED DESCRIPTION:
The purpose of this study is to adapt ESTEEM (Effective Skills to Empower Effective Men), developed by Dr. John Pachankis, to simultaneously target the multiple adverse health outcomes sexual minority women disproportionately face, including depression, suicidality, and alcohol abuse, that are linked to minority stress processes.

Project EQuIP will adapt the ESTEEM program for sexual minority women in three distinct phases. The focus of this registered protocol will be Phase 3, however Phases 1, 2 and 3 are described below.

Phase 1 will involve conducting interviews with 20 sexual minority women (SMW) who report experiencing depression, suicidality, and alcohol abuse. Information from these interviews will be used to gather insight from participants that can help inform the adaptation of a cognitive-behavioral treatment approach to specifically target sexual minority women's unique experiences with minority stress.

Phase 2 will involve consultation interviews with 10 community-based mental health experts who treat psychosocial health problems among at-risk SMW. Involvement of key community members in intervention design optimizes intervention dissemination and allows frontline professionals to shape the intervention that they would be most willing to implement. Input of mental health experts working with the SMW community will be used in order to translate existing, but largely untapped, clinical wisdom regarding SMW's minority stress experiences, mental health, and alcohol use into the development of the intervention.

Phase 3 will involve pilot testing the adapted cognitive-behavioral treatment through a randomized controlled trial with 60 SMW who report experiencing depression, anxiety, and alcohol abuse.

ELIGIBILITY:
For Phase 3

Inclusion Criteria:

* sexual minority status operationalized as identity (e.g., lesbian, bisexual, pansexual, queer)
* aged 18-35
* self-identification as a woman with the option of selecting multiple gender identities
* symptoms of anxiety or depression within the past 90 days (≥ 2.5 on the BSI-4 for either anxiety or depression)
* at least one instance of past-90-day heavy drinking (i.e., ≥ 4 drinks in one sitting)
* 6-month NYC residential stability and availability
* English fluency

Exclusion Criteria:

* active psychosis or active mania
* active suicidality or active homicidality
* currently in mental health treatment exceeding one day per month
* having received any cognitive-behavioral therapy treatment in the past 12 months
* evidence of gross cognitive impairment

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self- identification as a woman with the option of selecting multiple gender identities
Enrollment: 60 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pachankis, PhD, Principal Investigator — Associate Professor of Public Health (Social and Behavioral Sciences)
Locations (1):
- Yale LGBTQ+ Mental Health Initiative - Research Lab, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radloff, L. S. (1977). The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1, 385-401. http://dx.doi.org/10.1177/014662167700100306
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Alterman AI, Cacciola JS, Ivey MA, Habing B, Lynch KG. Reliability and validity of the alcohol short index of problems and a newly constructed drug short index of problems. J Stud Alcohol Drugs. 2009 Mar;70(2):304-7. doi: 10.15288/jsad.2009.70.304. PMID 19261243
- [Background] Bentley KH, Gallagher MW, Carl JR, Barlow DH. Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess. 2014 Sep;26(3):815-830. doi: 10.1037/a0036216. Epub 2014 Apr 7. PMID 24708078
- [Background] Norman SB, Cissell SH, Means-Christensen AJ, Stein MB. Development and validation of an Overall Anxiety Severity And Impairment Scale (OASIS). Depress Anxiety. 2006;23(4):245-9. doi: 10.1002/da.20182. PMID 16688739
- [Background] van Spijker BA, Batterham PJ, Calear AL, Farrer L, Christensen H, Reynolds J, Kerkhof AJ. The suicidal ideation attributes scale (SIDAS): Community-based validation study of a new scale for the measurement of suicidal ideation. Suicide Life Threat Behav. 2014 Aug;44(4):408-19. doi: 10.1111/sltb.12084. Epub 2014 Feb 24. PMID 24612048
- [Background] Dyar C, Feinstein BA, Eaton NR, London B. The Mediating Roles of Rejection Sensitivity and Proximal Stress in the Association Between Discrimination and Internalizing Symptoms Among Sexual Minority Women. Arch Sex Behav. 2018 Jan;47(1):205-218. doi: 10.1007/s10508-016-0869-1. Epub 2016 Oct 17. PMID 27752853
- [Background] Meyer IH, Rossano L, Ellis JM, Bradford J. A brief telephone interview to identify lesbian and bisexual women in random digit dialing sampling. J Sex Res. 2002 May;39(2):139-44. doi: 10.1080/00224490209552133. PMID 12476246
- [Background] Mohr JJ, Kendra MS. Revision and extension of a multidimensional measure of sexual minority identity: the Lesbian, Gay, and Bisexual Identity Scale. J Couns Psychol. 2011 Apr;58(2):234-245. doi: 10.1037/a0022858. PMID 21319899
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54. http:// dx.doi.org/10.1023/B:JOBA.0000007455.08539.94
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Treynor, W., Gonzalez, R., & Nolen-Hoeksema, S. (2003). Rumination reconsidered: A psychometric analysis. Cognitive Therapy and Re- search, 27, 247-259. http://dx.doi.org/10.1023/A:1023910315561
- [Background] Rathus, S. A. (1973). A 30-item schedule for assessing assertive behavior. Behavior Therapy, 4, 398-406. http://dx.doi.org/10.1016/S0005- 7894(73)80120-0
- [Result] Pachankis JE, McConocha EM, Clark KA, Wang K, Behari K, Fetzner BK, Brisbin CD, Scheer JR, Lehavot K. A transdiagnostic minority stress intervention for gender diverse sexual minority women's depression, anxiety, and unhealthy alcohol use: A randomized controlled trial. J Consult Clin Psychol. 2020 Jul;88(7):613-630. doi: 10.1037/ccp0000508. Epub 2020 May 21. PMID 32437174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapy | Waitlist
Started | 30 | 30
Three-month Pre-intervention | 0 (Participants in this arm started therapy immediately after randomization, and therefore, did not have a three-month waiting period prior to receiving the intervention.) | 30
Immediate Pre-intervention | 30 | 29
Post-intervention | 25 | 26
Three-month Follow-up (Post Intervention) | 25 | 0 (Participants in this arm started therapy three months after randomization (waitlist) and therefore, were not assessed at the three-month follow-up time point due to completion of the study)
Completed | 25 | 26
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapy | Waitlist | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.27 (3.35) | 25.90 (3.20) | 25.58 (3.26)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender women | 13 | 21 | 34
  Gender diverse (transgender, gender queer, nonbinary, gender fluid) | 17 | 9 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 22 | 19 | 41
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Sexual Orientation [Count of Participants; unit: Participants]
  Lesbian | 6 | 3 | 9
  Queer | 15 | 18 | 33
  Other (asexual, bisexual, pansexual, uncertain) | 9 | 9 | 18
Education level [Count of Participants; unit: Participants]
  Some college/currently in college | 5 | 8 | 13
  4-year college degree | 17 | 17 | 34
  Some graduate school or higher | 5 | 4 | 9
  Not reported | 3 | 1 | 4
Employment status [Count of Participants; unit: Participants]
  Full-time (40+ hours per week) | 18 | 15 | 33
  Part-time employment (<40 hours per week) | 8 | 8 | 16
  Student | 3 | 4 | 7
  Unemployed | 1 | 3 | 4
Personal Income, annually [Count of Participants; unit: Participants]
  Less than $29,000 | 15 | 17 | 32
  $30,000-49,999 | 10 | 2 | 12
  More than $50,000 | 5 | 11 | 16
Relationship status [Count of Participants; unit: Participants]
  Single or casually dating | 16 | 13 | 29
  Partnered | 13 | 17 | 30
  Not reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: The measure depression in participants, the Center for Epidemiological Studies - Depression Scale (CES-D) will be used. An overall depression score is computed as the sum of the 20 items, with Items 3, 11, 14, and 16 reversed. In cases with internally missing data (items not answered), the sums were computed after imputation of the missing values: # items on scale / # actually answered, multiplied by the sum obtained from the answered items. A higher score indicates more depressive symptomatology during the past week. Range is 0 - 60.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: Participants in the Therapy started therapy immediately after randomization, and therefore, have no data for the three-month waiting period prior to receiving the intervention. Participants in this arm started therapy three months after randomization (waitlist) and therefore, were not assessed at the three-month follow-up time point due to completion of the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 27.57 (1.80)
  Immediate Pre-intervention | 29.70 (1.84) | 26.86 (1.91)
  Post-intervention | 20.44 (1.80) | 24.83 (2.44)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 19.00 (2.18) |

2. Primary Outcome: Brief Symptom Inventory
Description: The Global Severity Index of the 18-item BSI provides a mean score across depression, anxiety, and somatization subscales, and assesses psychological distress (e.g., "feeling nervousness or shakiness inside") on a 5-point scale from 0 (not at all) to 4 (extremely) for the past 7 days. Scores range from 0-72, with higher scores indicating worse outcomes (greater symptoms severity).
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
units on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 1.80 (0.10)
  Immediate Pre-intervention | 1.74 (0.14) | 1.85 (0.09)
  Post-intervention | 1.38 (0.11) | 1.64 (0.11)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 1.16 (0.14) |

3. Primary Outcome: Alcohol Use
Description: Alcohol use will be measured using the Short Index of Problems for Alcohol (SIP-A). The SIP-A is a 15-item, binary response (yes/no) measure that has a range of scores from 0-15. The highest score of 15 is an indicator of the greatest amount of alcohol use related problems.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 3.93 (0.54)
  Immediate Pre-intervention | 3.63 (0.57) | 3.34 (0.60)
  Post-intervention | 2.16 (0.37) | 2.80 (0.64)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 1.92 (0.44) |

4. Secondary Outcome: Overall Depression Severity and Impairment Scale
Description: ODSIS is a 5-item scale that asks individuals to rate the severity and impairment associated with past-week symptoms of depression (e.g., "In the past week, when you have felt depressed, how intense or severe was your depression?) from 0 (little or none: Depression was absent or barely noticeable.) to 4 (extreme: Depression was overwhelming.). Scores range from 0-20, with higher scores indicating greater depression and associated impairment in the past week.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 6.17 (0.78)
  Immediate Pre-intervention | 6.30 (0.83) | 7.69 (0.73)
  Post-intervention | 4.09 (0.71) | 5.85 (0.82)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 3.88 (0.69) |

5. Secondary Outcome: Overall Anxiety Severity and Impairment Scale
Description: OASIS is a 5-item scale that asks individuals to rate the severity and impairment associated with past-week anxiety symptoms (e.g., "In the past week, when you have felt anxious, how intense or severe was your anxiety?") from 0 (little or none: Anxiety was absent or barely noticeable.) to 4 (extreme: Anxiety was overwhelming. It was impossible to relax at all. Physical symptoms were unbearable). Scores range from 0-20, with higher scores indicating greater anxiety and associated impairment in the past week.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 8.20 (0.46)
  Immediate Pre-intervention | 8.80 (0.64) | 8.03 (0.46)
  Post-intervention | 6.00 (0.70) | 6.08 (0.60)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 6.17 (0.68) |

6. Secondary Outcome: Suicidal Ideation Attributes Scale
Description: SIDAS is a 5-item scale that assesses past-month frequency and controllability of suicidal thoughts, how close one has come to making an attempt, and distress and impairment associated with thoughts of suicide (e.g., "In the past month, how often have you had thoughts about suicide?"). Responses range from 0 (never or not at all) to 10 (always or extremely) on each item, with item 2 reverse scored. Scale scores range from 0-50, with higher scores indicating more (worse) suicidal ideation.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 5.03 (1.42)
  Immediate Pre-intervention | 4.13 (1.51) | 5.59 (1.58)
  Post-intervention | 2.09 (1.04) | 2.73 (1.05)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 1.46 (0.75) |

7. Secondary Outcome: Lesbian, Gay, and Bisexual Identity Scale-Internalized Homonegativity Subscale
Description: Internalized stigma was assessed us- ing the mean score on a three-item scale, the Lesbian, Gay, and Bisexual Identity Scale-Internalized Homonegativity Subscale, that asks individuals to rate thoughts and feelings related to their LGBTQ identity (e.g., "If it were possible, I would choose to be straight"). Responses range from 1 (disagree strongly) to 6 (agree strongly). Scores range from 3-18 with higher scores indicating higher internalized stigma.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 1.49 (0.13)
  Immediate Pre-intervention | 1.72 (0.19) | 1.32 (0.10)
  Post-intervention | 1.63 (0.16) | 1.36 (0.12)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 1.49 (0.13) |

8. Post Hoc Outcome: Sexual Minority Women's Rejection Sensitivity Scale
Description: The Sexual Minority Women Rejection Sensitivity Scale asks participants to rate 16 vignettes in terms of how concerned or anxious each would make them about being rejected because of their sexual orientation, and their likelihood of attributing the rejection to their sexual orientation. For example, one item states, "You are on a date with a woman at a restaurant. Your waiter provides you and your date with poor service." Responses to the anxiety and likelihood stems range from 1 (very unconcerned/very unlikely) to 7 (very concerned/very likely). Total score is the sum of the products of anxiety and likelihood scores for all items. We adapted the scale to indicate "woman, gender nonconforming, or non-binary partner" and "heterosexual, cisgender" as relevant. Scale scores range from 16-112, with higher scores indicating higher rejection sensitivity.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 24.98 (1.63)
  Immediate Pre-intervention | 25.19 (1.38) | 23.03 (1.58)
  Post-intervention | 22.10 (1.51) | 22.12 (1.76)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 22.78 (1.72) |

9. Post Hoc Outcome: Sexual Orientation Concealment
Description: In the Sexual Orientation Concealment Scale, participants rate the degree to which they have disclosed their sexual orientation on a scale from 1 (out to none) to 4 (out to all). The total score is the mean of responses in the following domains: "family," "LGBTQ friends," "straight, cisgender friends," "co- workers", and "health care providers." Scores range from 1-4 with higher scores indicating lower sexual orientation concealment.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 1.89 (0.12)
  Immediate Pre-intervention | 1.87 (0.11) | 1.67 (0.12)
  Post-intervention | 1.74 (0.12) | 1.77 (0.14)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 1.75 (0.13) |

10. Post Hoc Outcome: Difficulties in Emotion Regulation Scale-Short Form
Description: In the Difficulties in Emotion Regulation Scale-Short Form (DERS- SF), an 18-item scale, individuals are asked how much each statement regarding emotion regulation (e.g., "When I'm upset, I acknowledge my emotions") applies to them from 1 (almost never) to 5 (almost always). Scores range from 18-90 with higher scores indicating greater difficulties in emotion regulation.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 49.37 (1.92)
  Immediate Pre-intervention | 47.50 (1.82) | 47.07 (1.74)
  Post-intervention | 40.74 (1.89) | 45.85 (1.72)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 40.58 (1.64) |

11. Post Hoc Outcome: Multidimensional Scale of Perceived Social Support
Description: The mean score on the Multidimensional Scale of Perceived Social Support (MSPSS), a 12-item scale, indicates the perceived support that individuals report receiving from family (e.g., "My family really tries to help me"), friends (e.g., "I have friends with whom I can share my joys and sorrows"), and significant others (e.g., "I have a special person who is a real source of comfort to me") on a scale ranging from 0 (very strongly disagree) to 7 (very strongly agree). Scores range from 0-72 with higher scores indicating greater perceived social support.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 3.39 (0.25)
  Immediate Pre-intervention | 3.72 (0.21) | 5.39 (0.14)
  Post-intervention | 4.31 (0.28) | 5.35 (0.17)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 5.12 (0.24) |

12. Post Hoc Outcome: Ruminative Responses Scale-Brooding Subscale
Description: The sum of the five items on the Ruminative Responses Scale- Brooding Subscale (RRS) indicates the frequency with which participants experience brooding thoughts in response to depressed mood (e.g., "Think 'what am I doing to deserve this?'") along a scale ranging from 1 (almost never) to 4 (almost always). Scores range from 5-20 with higher scores indicating greater rumination.
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 13.57 (0.55)
  Immediate Pre-intervention | 13.80 (0.45) | 13.52 (0.54)
  Post-intervention | 12.91 (0.57) | 12.04 (0.66)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 11.25 (0.48) |

13. Post Hoc Outcome: Simple Rathus Assertiveness Schedule-Short Form
Description: The Simple Rathus Assertiveness Schedule-Short Form (SRAS-SF), a 19-item scale, asks individuals to rate the personal typicality of assertive and unassertive behavior (e.g., "I find it embarrassing to return merchandise," "I have avoided asking questions for fear of sounding stupid") along a scale from 1 (very uncharacteristic of me) to 6 (very characteristic of me), for a summed total score.
  Scores range from 19-114 with higher scores indicating greater unassertiveness (scale was reverse-scored).
Time Frame: Three-month pre-intervention, Immediate Pre-intervention, Post-intervention, Three-month Follow-up (Post Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapy | Waitlist
Number analyzed (Participants) | 30 | 30
score on a scale
  Three-month pre-intervention: number analyzed (Participants) | 0 | 30
  Three-month pre-intervention |  | 62.80 (2.67)
  Immediate Pre-intervention | 66.87 (3.10) | 57.86 (2.11)
  Post-intervention | 62.43 (3.05) | 59.42 (2.29)
  Three-month Follow-up (Post Intervention): number analyzed (Participants) | 30 | 0
  Three-month Follow-up (Post Intervention) | 62.46 (3.13) |

ADVERSE EVENTS:
Time Frame: From baseline through study completion (up to 6 months).
Description: Participants' risk for suicide was assessed at baseline, 3-month follow-up and 6-month follow-up assessments using the Brief Symptom Inventory and Suicidal Ideation Attributes Scale, and through participant self-disclosure (e.g., during therapy). Participants randomized to waitlist were assessed for the 3-month waiting period, and then assessed while in therapy for the 3-month period. Participants randomized to immediate therapy were assessed for adverse events for the full 6 months.
Groups:
- Therapy: Individuals assigned to therapy will receive 10 weekly individually-delivered sessions, directly after randomization, that address minority stress mechanisms underlying SMW's depression, anxiety, and alcohol abuse.
  EQuIP (Empowering Queer Identities in Psychotherapy): Individuals assigned to therapy will receive 10 weekly individually-delivered sessions, directly after baseline assessment, that address minority stress mechanisms underlying SMW's depression, anxiety, and alcohol abuse.
- Waitlist: Individuals assigned to waitlist will be put on a waitlist for 3 months after randomization, after which they will also receive the same treatment as the therapy group.
Arm/Group | Therapy | Waitlist
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/30
Other Adverse Events (participants affected / at risk) | 0/60 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapy (N=60) | Waitlist (N=30)
Active suicidality (Psychiatric disorders) | 1 (1) | 0 (0) — Adverse event occurred during the intervention (therapy) phase of the waitlist arm of the study. The sample size for risk for adverse events under therapy reflects adverse events that occurred when participants were receiving the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03721276/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03721276/SAP_001.pdf
  • Informed Consent Form (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT03721276/ICF_002.pdf